CLINICAL TRIAL: NCT05523414
Title: A Pilot Feasibility Study to Evaluate the Effect of SKY Breath Meditation on Health and Well-being
Brief Title: The Effect of SKY Breath Meditation on Health and Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Ritu Aneja, Professor and Associate Dean for Research & Innovation, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB-300009383
Record Dates: First submitted 2022-08-19; First posted 2022-08-31 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2024-04

CONDITIONS: Stress; Stress, Psychological; Stress, Physiological; Anxiety; Mental Well Being; Happiness; Resilience
Keywords: mindfulness; breathing; meditation; stress reduction; anxiety; depression; DNA methylation; epigenetic; wearable devices; heart rate variability
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders; Psychological Well-Being; Respiratory Aspiration; Depression

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either the SKY arm or the control arm, that practices the HEP.
Who Masked: Investigator
Masking Description: Only the Principal investigator and study coordinator will have access to identifying information. They will de-identify the data and then send this de-identified data (sequencing data and the other clinical, demographic and behavioral data) into an easily accessible set of files for further analysis by the remaining team members. They will also make sure there are no medical record numbers, intervention type, or other identifying information in this dataset, and that the data is blinded in this respect. The files will be stored behind a secure firewall, so that it can only be accessed with permission by the members of the study group. The data will denote the SKY and control groups as Arm 1 & Arm 2 without indicating whether they refer to SKY or the control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SKY (Experimental): In-person SKY sessions will be 3 hours long on each of 3 consecutive days, and participants must be willing to attend all 3 sessions. Each session comprises a combination of breathwork, emotional resilience training, yoga, and leadership skills. The SKY technique includes a unique set of standardized breathing techniques to rapidly reduce neuroendocrine stress responses and the autonomic imbalance due to sympathetic overdrive. 8 weeks of online and/or in-person sessions will be delivered to participants in the follow-up period after the initial in-person intervention. They will receive intermittent reminders about their daily practice during the 8-week follow-up period. The participants will be asked to engage in daily 30 minute SKY sessions remotely, that is led by an instructor. Each participant will be required to log in the number of times a week they practice. In addition, weekly 60-minute reinforcement sessions will be conducted, in-person.
  Interventions: Behavioral: SKY
- Control (No Intervention): Waitlist control participants will not be provided any intervention. However, they will have the same schedule for data and biological specimen collection as the SKY intervention participants. They will be provided an opportunity to take the SKY retreat free of charge at the end of the follow up period.

INTERVENTIONS:
Behavioral: SKY — The SKY intervention will be administered in-person over three sessions spread over three consecutive days by qualified instructors. Participants will then be followed up over eight weeks' time, where they will be given the option to attend daily 35 minute breathwork sessions, again, guided by experienced instructors. Participants will be required to log whether or not they practiced for each day in the eight-week period. They will also receive intermittent reminders about their daily practice during the 8-week follow-up period.
  Other Names: Sudarshan Kriya Yoga; SKY Breath Meditation
  Arms: SKY

SUMMARY:
The goal of this pilot SKY (Sudarshan Kriya Yoga) Breath Meditation study is to establish feasibility and acceptability of the intervention; and investigate preliminary effectiveness of the intervention at the DNA methylation, RNA and protein levels in blood samples collected from participants before and after the 8 week SKY intervention. Primary outcomes also include preliminary effectiveness at the physiological level using a wearable device used for continuous monitoring. Secondary outcome measures include behavioral inventories.

DETAILED DESCRIPTION:
The present study will recruit up to 60 participants in the SKY intervention and up to 60 participants in the control group. Recruitment is expected to take up to a year. After providing informed consent, participants will be randomly assigned to the SKY intervention group, or a waitlist control group. Interventions will be performed in-person in San Diego.

Prior to interventions, each participant will be asked to fill out behavioral questionnaires containing surveys and standardized cognitive measurements. Participants will be also asked to provide blood samples for biological assays (epigenetics, transcriptomics and proteomics). All participants will be scheduled for the questionnaire data collection and specimen collection up to two weeks preceding the start of either intervention. Participants will be asked to wear a Garmin vivoSmart5 smartwatch to collect physiological measures.

The SKY intervention will be administered in-person over three sessions over three consecutive days. All participants (SKY and control) will be asked to provide a second blood sample at the end of the third session of the SKY intervention. SKY participants will then engage in a remotely administered follow-up over up to eight weeks' time with the option to attend daily remotely-led breathwork sessions for 30 minutes. Participants will be asked to log daily practice engagement using online surveys through the eight-week follow-up period. Reminders will be provided to the participant intermittently during this time. During the period of eight weeks, the participants will return for 1-hour in-person follow-up SKY sessions once a week. They will be required to attend at least 75% of these weekly sessions. After 8 weeks of follow up, participants will provide a third sample of blood, and perform a post-intervention questionnaire.

Control participants will also have a similar schedule of data and biological sample collection as the SKY group. Waitlist controls will be provided the opportunity to attend the SKY retreat free of charge at the conclusion of the follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers over 21 years of age who are willing to meet the standards of the study.
* Minimum 5th grade equivalent competency in English
* Agree to complete all follow up sessions per week of SKY Breath practice.

Exclusion Criteria:

* Diagnosis of any major medical condition including, but not limited to: dementia, severe hypertension, cancer, diabetes, rheumatoid arthritis, asthma or respiratory illnesses, history of seizure disorder, Crohn's disease, lupus, colitis, dermatitis, fibromyalgia, HIV, hepatitis B or C.
* Diagnosis of any psychiatric condition including, but not limited to: severe clinical depression, bipolar disorder, schizophrenia/schizoaffective disorder, suicidal ideation, ADHD
* Recent history of major psychotic episode within the last 12 months
* Recent history of consistent substance dependence or abuse either by history or self-report within the last 3 months
* Major surgery within last 12 weeks
* On hormone-replacement therapy
* Taking lithium or lithium-based medication
* Currently pregnant/breastfeeding or actively trying to become pregnant
* BMI greater than 35
* Exhibiting symptoms like prolonged cognitive fog or difficulty breathing.
* Smokes any tobacco products (including cigarettes, vapes, hookah)
* Heavy alcohol drinker (per CDC definition, 8 or more drinks per week for women, 15 or more drinks per week for men)
* Concurrently participating in another pilot study/clinical trial of a mind/body intervention
* Regularly practices (3+ times a week) a formal meditation or breath-based technique

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Up to 1 year
  Descriptive statistics will be used to compute the proportion of screen-eligible participants enrolled by consent. Proportions will be computed, along with 95% confidence intervals, to indicate the precision of the point estimate.
Refusal rate | Up to 1 year
  Descriptive statistics will be used to compute the proportion of screen-eligible individuals who refused to participate. Proportions will be computed, along with 95% confidence intervals, to indicate the precision of the point estimate.
Retention rate | Week to week during 8 weeks
  Among the participants who originally attended the 3-day workshop, descriptive statistics will be used to compute proportion of participants that complete all 8 SKY follow-up study visits. Proportions will be computed, along with 95% confidence intervals, to indicate the precision of the point estimate.
Adherence rate | 8 weeks during intervention period
  Descriptive statistics will be used to compute the frequency of home practice completion, weekly, by the intervention participants. Proportions will be computed, along with 95% confidence intervals, to indicate the precision of the point estimate.
Heart rate variability | Continuous monitoring over 8-week intervention
  Heart rate variability will be collected using the Garmin vivosmart5 watch
Respiration rate | Continuous monitoring over 8-week intervention
  Respiration rate will be measured using the Garmin vivosmart5 watch

SECONDARY OUTCOMES:
Perceived Stress Scale | Pre/post 8-week intervention
  The Perceived Stress Scale (PSS) is the most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. Lower values indicate less stress.
Brief-COPE | Pre/post 8-week intervention
  The Brief-COPE is a 28 item self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event. Higher scores indicate difficulty with coping.
Pittsburgh Sleep Quality Assessment | Pre/post 8-week intervention
  The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the last month. Higher scores indicate more sleep disturbances.
Mini-Mood and Anxiety Symptom Questionnaire | Pre/post 8-week intervention
  The Mood and Anxiety Symptom Questionnaire (MASQ) is an instrument containing a range of symptoms relevant to depression and anxiety. Items are evaluated for Distress, Anxiety, Depression with higher scores on subcomponents indicate more extreme levels of each metric.
SF-12v2 | Pre/post 8-week intervention
  The SF-12v2 is a health-related quality-of-life questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health. Higher scores indicate better physical and mental health.
Social-Connectedness Scale | Pre/post 8-week intervention
  The social connectedness scale assesses the degree to which persons feel connected to others in their social environment. Higher scores indicate more social connectedness. The Social Connectedness Scale Revised [SCS-R; Cronbach's Alpha=0.94] will be used to measure social connectedness.
Epigenetic (DNA Methylation) changes | Pre/post 8 week intervention, and Day 3 (midpoint)
  DNA Methylation changes in SKY and control groups (pre vs post interventions) will be measured by EPIC v2 array and whole-genome bisulfite sequencing (WGBS). Data analyses will be performed utilizing previously published standard pipelines.
Gene expression changes | Pre/post 8 week intervention, and Day 3 (midpoint)
  RNA level changes between SKY and control groups will be examined.
Proteomic changes | Pre/post 8 week intervention
  Protein level changes between SKY and control groups will be examined.

OTHER OUTCOMES:
Cytokine changes in serum samples | Pre/post 8-week intervention
  Cytokine changes will be measured using ELISA assay on the blood sample collected and a standard ELISA panel for pro-inflammatory cytokines will be used to detect changes in their levels post intervention.
Assessment of changes in mitochondrial DNA damage-associated molecular patterns (mtDNA DAMPs) from blood serum. | Pre/post 8-week intervention
  Cell-free DNA will be eluted to a specified serum volume and used for the mtDNA DAMPs assays.
Serum biomarkers | Pre/post 8-week intervention
  Serum samples will be collected using standard procedures from the blood samples and immunoassayed using enzyme-linked immunosorbent assay to detect serum biomarkers

CONTACTS AND LOCATIONS:
Locations (1):
- Study Site: Confidential, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No